CLINICAL TRIAL: NCT00233545
Title: Miltefosine to Treat Cutaneous Leishmaniasis in Bolivia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-2005
Record Dates: First submitted 2005-09-28; First posted 2005-10-06 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Cutaneous Leishmaniasis
Keywords: cutaneous; leishmaniasis; drug; miltefosine
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — miltefosine; Antimony

INTERVENTIONS:
Drug: miltefosine
Drug: antimony

SUMMARY:
Cutaneous leishmaniasis is typically treated with the parenteral product pentavalent antimony. Miltefosine is an oral agent shown to be active for mucosal leishmaniasis due to L braziliensis in Bolivia and cutaneous leishmaniasis due to L panamensis in Colombia. This trial is intended to evaluate miltefosine for cutaneous leishmaniasis due to L braziliensis in Bolivia. Patients will be randomly assigned to miltefosine or pentavalent antimony. Standard dose regimens will be used for both drugs.

ELIGIBILITY:
Presentation: At least 1 lesion must be ulcerative. Parasitology: Parasitological confirmation of 1 lesion will be made by visualization or culture of leishmania from the biopsy or aspirate of the lesion.

Previous RX: No specific or putatively specific therapy for leishmaniasis (Sb, pentamidine, amphotericin B, imidazoles, allopurinol)

Other diseases: No concomitant diseases by history and by approximately normal complete blood counts (white blood count, hemoglobin, platelet count), values of liver transaminases (SGOT) and kidney function tests (creatinine).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2005-09; Study Completion 2007-09

PRIMARY OUTCOMES:
cure rate

CONTACTS AND LOCATIONS:
Overall Officials: J Soto, MD, Principal Investigator — FADER
Locations (1):
- Puesto de Salud, Campamento OSCAR,, Palos Blancos, Bolivia